CLINICAL TRIAL: NCT03616535
Title: Hemodialysis-based Interventions to Preserve Cognitive Function
Brief Title: Interventions Made to Preserve Cognitive Function
Acronym: IMPCT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: DSMB terminated study due to COVID-19 delays in recruitment
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: IRB00152858; R01DK114074 (NIH)
Record Dates: First submitted 2018-06-13; First posted 2018-08-06 (Actual); Results first posted 2025-04-11 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-06

CONDITIONS: ESRD
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Cognitive Training; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cognitive training (Active Comparator): Participants randomized to CT will play "brain games" on a tablet. They will be asked to engage in the activity for a minimum of 30 minutes during each hemodialysis session for 6 months. At each HD session, participants will have 10 different brain games to play and the games will vary for each session.
  Interventions: Other: Cognitive training
- Exercise training (Active Comparator): Participants randomized to the ET arm will be given a stationary foot peddler and will be asked to engage in the activity for a minimum of 30 minutes at each hemodialysis session for 6 months. ET will start with a 2 minute warm up, then the resistance will be adjusted so that participants are working at perceived exertion of "somewhat strong," using the Borg scale (87) (~50 rpm). Resistance will be increased when the rating falls below "somewhat hard."
  Interventions: Other: Exercise training
- Combined cognitive and exercise training (Active Comparator): Participants in the CT+ET arm will start with 30 minutes of CT (playing "brain games" on tablet) with a 15-minute break, and then, 30 minutes of ET (stationary foot peddler).
  Interventions: Other: Combined cognitive and exercise training
- Standard of Care (No Intervention): Participants in this arm will receive standard of care

INTERVENTIONS:
Other: Cognitive training — The investigators will provide participants with tablets to play brain games.
  Other Names: CT
  Arms: Cognitive training
Other: Exercise training — The investigators will provide participants with foot peddlers.
  Other Names: ET
  Arms: Exercise training
Other: Combined cognitive and exercise training — The investigators will provide participants with tablets to play brain games for cognitive training and stationary foot peddlers for exercise training.
  Other Names: CT+ET
  Arms: Combined cognitive and exercise training

SUMMARY:
This is a randomized, controlled trial to slow cognitive decline in adults undergoing hemodialysis (HD). The investigators will test three interventions cognitive training (CT), exercise training (ET), and combined cognitive and exercise training (CT+ET) relative to standard of care (SC).

DETAILED DESCRIPTION:
This will be a two by two factorial, randomized, controlled trial to slow cognitive decline in adults undergoing hemodialysis (HD). The investigators primary objective is to determine if receiving cognitive training (tablet-based brain games), exercise training (stationary foot pedal), or combined cognitive and exercise training preserves executive function relative to those with standard of care . The secondary objectives are to compare the rates of end stage renal disease (ESRD)-specific clinical outcomes and patient centered outcomes among those receiving CT, or ET, or CT+ET relative to those in SC. The investigators will formally test whether receiving CT or ET will preserve executive function and receiving combined CT+ET will preserve executive function better than CT or ET alone.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older at enrollment
* English speaking
* within 3 months to 3 years of initiating hemodialysis
* receiving hemodialysis at participating dialysis centers

Exclusion Criteria: Patients with the following conditions will be excluded:

* Pregnancy
* Angina Pectoris
* Chronic lung disease requiring oxygen
* Musculoskeletal conditions that limit mobility
* Upper or lower extremity amputation
* Orthopedic disorders exacerbated by physical activity
* Femoral arteriovenous (AV) access
* Hepatitis B infection
* Blindness/Legal blindness

In addition to conditions outlined above, patients who are currently incarcerated will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2018-08-30 (Actual); Primary Completion 2023-06-23 (Actual); Study Completion 2023-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aarti Mathur, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins School of Medicine, Baltimore, Maryland
  - New York University Langone Health, New York, New York

REFERENCES:
- [Derived] Bernier-Jean A, Beruni NA, Bondonno NP, Williams G, Teixeira-Pinto A, Craig JC, Wong G. Exercise training for adults undergoing maintenance dialysis. Cochrane Database Syst Rev. 2022 Jan 12;1(1):CD014653. doi: 10.1002/14651858.CD014653. PMID 35018639
- [Derived] McAdams-DeMarco MA, Chu NM, Steckel M, Kunwar S, Gonzalez Fernandez M, Carlson MC, Fine DM, Appel LJ, Diener-West M, Segev DL. Interventions Made to Preserve Cognitive Function Trial (IMPCT) study protocol: a multi-dialysis center 2x2 factorial randomized controlled trial of intradialytic cognitive and exercise training to preserve cognitive function. BMC Nephrol. 2020 Sep 3;21(1):383. doi: 10.1186/s12882-020-02041-y. PMID 32883245

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was stopped after enrolling 130 participants by the Data Safety Monitoring Board (DSMB) due to COVID-19 shutdowns.
Pre-assignment Details: 130 participants were consented. There were 9 participants who were consented but not randomized due to COVID-19 shutdowns. They are not included in the results.
Groups:
- Cognitive Training: Participants randomized to CT will play "brain games" on a tablet. They will be asked to engage in the activity for a minimum of 30 minutes during each hemodialysis (HD) session. At each HD session, participants will have 10 different brain games to play and the games will vary for each session.
  Cognitive training: The investigators will provide participants with tablets to play brain games.
- Exercise Training: Participants randomized to the Exercise Training (ET) arm will be given a stationary foot peddler and will be asked to engage in the activity for a minimum of 30 minutes at each hemodialysis session. ET will start with a 2 minute warm up, then the resistance will be adjusted so that participants are working at perceived exertion of "somewhat strong," using the Borg scale (87) (~50 rpm). Resistance will be increased when the rating falls below "somewhat hard."
  Exercise training: The investigators will provide participants with foot peddlers.
Period: Overall Study
Arm/Group | Cognitive Training | Exercise Training | Combined Cognitive and Exercise Training | Standard of Care
Started | 31 | 29 | 35 | 26
Completed | 24 | 23 | 27 | 21
Not Completed | 7 | 6 | 8 | 5
Not completed — Death | 2 | 0 | 0 | 1
Not completed — Lost to Follow-up | 2 | 1 | 0 | 2
Not completed — Withdrawal by Subject | 1 | 2 | 5 | 1
Not completed — Not specified or change in eligibility | 2 | 3 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Cognitive Training: Participants randomized to CT will play "brain games" on a tablet. They will be asked to engage in the activity for a minimum of 30 minutes during each hemodialysis session. At each HD session, participants will have 10 different brain games to play and the games will vary for each session.
  Cognitive training: The investigators will provide participants with tablets to play brain games.
- Exercise Training: Participants randomized to the ET arm will be given a stationary foot peddler and will be asked to engage in the activity for a minimum of 30 minutes at each hemodialysis session . ET will start with a 2 minute warm up, then the resistance will be adjusted so that participants are working at perceived exertion of "somewhat strong," using the Borg scale (87) (~50 rpm). Resistance will be increased when the rating falls below "somewhat hard."
  Exercise training: The investigators will provide participants with foot peddlers.
- Total: Total of all reporting groups
Arm/Group | Cognitive Training | Exercise Training | Combined Cognitive and Exercise Training | Standard of Care | Total
Number analyzed (Participants) | 31 | 29 | 35 | 26 | 121
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 64.2 [56.2 to 69.9] | 58.4 [48.9 to 66.0] | 60.4 [52.0 to 70.3] | 60.4 [38.3 to 66.5] | 61.5 [52.0 to 67.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 14 | 10 | 45
  Male | 20 | 19 | 21 | 16 | 76
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 5 | 7 | 9 | 6 | 27
  Black/African American | 25 | 22 | 23 | 19 | 89
  Asian/Asian American | 1 | 0 | 3 | 1 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 31 | 29 | 35 | 26 | 121

OUTCOME MEASURES:

1. Primary Outcome: Change in Executive Function as Assessed by the Trail Making Test Assessment (TMT)
Description: Change in executive function between baseline and 3 months as assessed by the Trail Making Test which is comprised of Part A and Part B. Executive function is assessed by the time (seconds) to complete Part B minus the time (seconds) to complete Part A. Needing more time to complete the test indicates worse executive function.
Time Frame: 3 months
Population: Due to COVID-19 shutdowns, the trial was terminated early by the DSMB. All participants with available TMT A/B at baseline and 3 months of follow-up were analyzed.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Cognitive Training | Exercise Training | Combined Cognitive and Exercise Training | Standard of Care
Number analyzed (Participants) | 24 | 23 | 27 | 21
seconds | 20.4 (54.9) | -0.8 (82) | -5.6 (101.7) | 5.7 (53.2)

2. Secondary Outcome: Change in Global Cognitive Function as Measured by the Montreal Cognitive Assessment (MoCA)
Description: Change in global cognitive function at 3-months of interventions as measured by the Montreal Cognitive Assessment (MoCA). It is a brief 30 question test that assesses different cognitive domains: attention and concentration, executive functions, memory, language, visual construction skills, conceptual thinking, calculations, and orientation. Total possible score range is 0-30 points, and a score of 26 or above is considered normal.
Time Frame: Baseline, 3 months
Population: Participants with an available MoCA at baseline and 3-month follow-up were included in this analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Training | Exercise Training | Combined Cognitive and Exercise Training | Standard of Care
Number analyzed (Participants) | 20 | 17 | 22 | 18
score on a scale | -0.1 (2.9) | 0.1 (2.1) | 1.5 (3.1) | -0.6 (3.3)

3. Secondary Outcome: Number of Participants Completing Executive Function as Measured by the Stroop Test
Description: Number completing the Stroop test of executive function at 3 months of interventions. The Stroop test asks participants to view two conflicting pieces of information, specifically the word itself and the color of the ink it's printed in. Participants are asked to name the color of the ink used to print words, rather than reading the words themselves.
Time Frame: 3 months
Population: Participants with an available Stroop test at 3-month follow-up were included in this analysis.
Measure: Number; unit: participants
Arm/Group | Cognitive Training | Exercise Training | Combined Cognitive and Exercise Training | Standard of Care
Number analyzed (Participants) | 16 | 16 | 22 | 14
participants | 16 | 14 | 19 | 13

4. Secondary Outcome: Change in Executive Function as Measured by the Digit Symbol Substitution Test
Description: Change in executive function at 3 months of interventions as measure by the Digit Symbol Substitution Test. This test evaluates the speed and working memory components of executive function. It involves a key consisting of the numbers 1-9, each paired with a unique, easy-to--draw symbol such as a "V", "+" or ">". Below the key are a series of the numbers 1-9 in random order and repeated several times. The participant is allowed 90 seconds to fill in the corresponding symbol for each number. This task requires the individual to visually scan the answer key provided at the top of the test and then write the correct symbol by each number as quickly as possible. The correct number of symbols written within 90 seconds is measured. Total possible score ranges from a minimum of 0 to a maximum of 90 points. Higher scores represent better outcomes.
Time Frame: baseline and 3 months
Population: Participants with an available Digit Symbol Substitution Test at baseline and 3-month follow-up were included in this analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Training | Exercise Training | Combined Cognitive and Exercise Training | Standard of Care
Number analyzed (Participants) | 20 | 19 | 23 | 15
score on a scale | 3.6 (12.8) | 6.4 (15.6) | 2.0 (18.9) | .7 (20)

5. Secondary Outcome: Change in Physical Function as Measured by the Short Physical Performance Battery (SPPB) Test
Description: Change in lower extremity function at 3 months of interventions using the SPPB test. The SPPB is an objective assessment tool for evaluating lower extremity functioning This test is a performance-based assessment comprised of 3 tasks: 1) repeated chair stands, 2) standing balance, and 3) a 4-meter usual paced walk in those with and without a walking aid (meters/second). Participants receive a score of 0 for a task if they were unable to complete the task; otherwise, they receive scores of 1-4 based on population-based norms. The scores of the three tasks are summed to create the SPPB score. The SPPB score ranges from 0 to 12, with lower scores indicating poorer function.
Time Frame: Baseline and 3 months
Population: Participants with an available SPPB at baseline and 3-month follow-up were included in this analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Training | Exercise Training | Combined Cognitive and Exercise Training | Standard of Care
Number analyzed (Participants) | 22 | 18 | 25 | 16
score on a scale | -1.5 (3.9) | -1.7 (3.8) | -0.1 (2.8) | 0.1 (1.8)

6. Secondary Outcome: Number of Participants With an Injurious Fall
Description: Number of participants with an injurious falls resulting in a medical encounter during the 6 months of interventions and for 6 months after the interventions
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cognitive Training | Exercise Training | Combined Cognitive and Exercise Training | Standard of Care
Number analyzed (Participants) | 31 | 29 | 35 | 26
Participants | 0 | 1 | 0 | 0

7. Secondary Outcome: Number of Participants With a Hospitalizations
Description: The number of participants with a hospitalizations during the 6 months of interventions and 6 months after the interventions
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cognitive Training | Exercise Training | Combined Cognitive and Exercise Training | Standard of Care
Number analyzed (Participants) | 31 | 29 | 35 | 26
Participants | 12 | 7 | 11 | 7

8. Secondary Outcome: Mortality
Description: Mortality will be ascertained within the 6 months of the intervention and 1 year after the intervention (1.5 years total).
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cognitive Training | Exercise Training | Combined Cognitive and Exercise Training | Standard of Care
Number analyzed (Participants) | 31 | 29 | 35 | 26
Participants | 6 | 4 | 3 | 4

9. Secondary Outcome: Change in Patient-centered Outcomes as Measured by the Kidney Disease Quality of Life (KDQOL) Survey
Description: Change in kidney disease-specific physical and mental quality of life at 3 months. Using a single the question from the KDQOL: In general, would you say your health is ___ ? It is reported on a 5-point score: 1, poor; 2, fair; 3, good; 4, very good; 5, excellent. Higher is better. While the score of KDQOL ranges from 1 to 5 points, we are measuring the 3-month change in this score. Therefore, the change could range from -4 to 4 points.
Time Frame: Baseline and 3 months
Population: Participants with available KDQOL at baseline and 3-month follow-up were included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Training | Exercise Training | Combined Cognitive and Exercise Training | Standard of Care
Number analyzed (Participants) | 23 | 21 | 28 | 18
units on a scale | -0.1 (1.1) | 0.2 (1.1) | 0.2 (0.7) | 0.3 (1.0)

10. Secondary Outcome: Change in Patient-centered Outcomes as Measured by the Patient-Reported Outcomes Measurement Information System (PROMIS)-29
Description: Change in Patient-centered Outcomes as measured by the Patient-Reported Outcomes Measurement Information System (PROMIS)-29 The change in PROMIS-29 score at 3 months is reported. Scores range from 0-140; higher scores are better.
Time Frame: Baseline and 3 months
Population: Only participants with available PROMIS-29 at baseline and 3 months were included.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Training | Exercise Training | Combined Cognitive and Exercise Training | Standard of Care
Number analyzed (Participants) | 23 | 21 | 27 | 18
score on a scale | 7.3 (22.2) | -0.4 (13.5) | -3.9 (19.8) | -5.6 (17.2)

11. Secondary Outcome: Number of Participants With an Amputation
Description: The number of participants with an amputation during the 6 months of interventions and 6 months after interventions. This information will be either self-reported by the participant or abstracted from the medical records to see if the interventions are associated with amputations
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cognitive Training | Exercise Training | Combined Cognitive and Exercise Training | Standard of Care
Number analyzed (Participants) | 31 | 29 | 35 | 26
Participants | 0 | 0 | 0 | 0

12. Secondary Outcome: Number of Participants Able to Return to Work
Description: The number of participants able to return to work during the 6 months of interventions and 6 months after interventions.
Time Frame: 12 months
Population: Among those who were unemployed or on leave of absence at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Cognitive Training | Exercise Training | Combined Cognitive and Exercise Training | Standard of Care
Number analyzed (Participants) | 3 | 4 | 8 | 3
Participants | 1 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 18 months after enrollment for mortality; up to 12 months after enrollment for hospitalizations; all else up to 6 months.
Groups:
- Exercise Training: Participants randomized to the ET arm will be given a stationary foot peddler and will be asked to engage in the activity for a minimum of 30 minutes at each hemodialysis session. ET will start with a 2 minute warm up, then the resistance will be adjusted so that participants are working at perceived exertion of "somewhat strong," using the Borg scale (87) (~50 rpm). Resistance will be increased when the rating falls below "somewhat hard."
  Exercise training: The investigators will provide participants with foot peddlers.
Arm/Group | Cognitive Training | Exercise Training | Combined Cognitive and Exercise Training | Standard of Care
All-Cause Mortality (participants affected / at risk) | 6/31 | 4/29 | 3/35 | 4/26
Serious Adverse Events (participants affected / at risk) | 6/31 | 1/29 | 4/35 | 0/26
Other Adverse Events (participants affected / at risk) | 24/31 | 21/29 | 28/35 | 12/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cognitive Training (N=31) | Exercise Training (N=29) | Combined Cognitive and Exercise Training (N=35) | Standard of Care (N=26)
Hospitalization/Prolonged Hospitalization (General disorders) | 6 | 1 | 4 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cognitive Training (N=31) | Exercise Training (N=29) | Combined Cognitive and Exercise Training (N=35) | Standard of Care (N=26)
Cramp (Musculoskeletal and connective tissue disorders) | 14 | 13 | 15 | 7
Hypotension (General disorders) | 7 | 11 | 17 | 0
Hypertension (General disorders) | 12 | 10 | 10 | 4
Elevated heart rate (Cardiac disorders) | 0 | 3 | 3 | 0
headache (General disorders) | 6 | 7 | 13 | 4
other unexpected event (General disorders) | 14 | 7 | 13 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-18): https://cdn.clinicaltrials.gov/large-docs/35/NCT03616535/Prot_SAP_000.pdf